CLINICAL TRIAL: NCT05793788
Title: UCLA Health Patient Health Maintenance Outreach Text Message
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard K. Leuchter, MD, Clinical Instructor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MAPinitial
Record Dates: First submitted 2023-03-09; First posted 2023-03-31 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Health Maintenance; Diabetes; Cancer
Keywords: primary care; digital outreach
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel-arm randomized control trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Specific (Experimental): Eligible, randomized participant will receive a brief, specific SMS message informing patients that they should obtain screenings and tests they are due for.
  Interventions: Behavioral: Outreach Text Messages; Behavioral: Specific
- Arm 2: General (Experimental): Eligible, randomized participant will receive a brief, generic SMS message informing patients that they have a health gap to be closed.
  Interventions: Behavioral: Outreach Text Messages; Behavioral: General
- Arm 3: Intention-oriented; General (Experimental): Eligible, randomized participant will receive an intention-oriented, generic SMS message informing patients that they have a health gap to be closed and highlighting the importance of doing so.
  Interventions: Behavioral: Outreach Text Messages; Behavioral: General; Behavioral: Elevating Intentions
- Arm 4: Action-oriented; General (Experimental): Eligible, randomized participant will receive an action-oriented, generic SMS-message informing patients that they have a health gap to be closed and prompting them to act soon before they forget.
  Interventions: Behavioral: Outreach Text Messages; Behavioral: General; Behavioral: Prompting Action

INTERVENTIONS:
Behavioral: Outreach Text Messages — The investigators will send randomized participants an SMS message encouraging them to click provided link and close their outstanding, overdue preventive care measures.
  The provided link will take them to their MyChart login page; after logging in, they would see their personalized My Action Plan Letter detailing their personalized, overdue preventive care measures. Message content will vary based on randomization arm as noted below.
Behavioral: Specific — The message will inform patients that the care team has identified tests/screenings that they are due for.
  Arms: Arm 1: Specific
Behavioral: General — The message will inform patients that the care team has identified a care gap in their record.
  Arms: Arm 2: General; Arm 3: Intention-oriented; General; Arm 4: Action-oriented; General
Behavioral: Elevating Intentions — The message will point out that even if patients feel healthy, their doctor recommends them to take care of their health gaps.
  Arms: Arm 3: Intention-oriented; General
Behavioral: Prompting Action — The message will prompt patients to take care of their health gaps right away before they forget.
  Arms: Arm 4: Action-oriented; General

SUMMARY:
This is a prospective randomized clinical trial evaluating how behaviorally-informed outreach text messages impact patient engagement with primary care. This prospective randomized control trial is being implemented in conjunction with UCLA Health's larger quality improvement initiative (the My Action Plan Quality Improvement Initiative) in order to improve primary care preventive measure completion rates.

DETAILED DESCRIPTION:
Health maintenance measures have been shown to be critical in early detection, secondary prevention, and early management of numerous medical conditions--from diabetes to various cancers. The standardization of these health maintenance measures have resulted in major improvements in population health. Despite the importance of these primary care tests and screenings, many patients are overdue for these tests.

Given this healthcare gap, it is critical to investigate more effective strategies to facilitate health maintenance measure completion. This study aims to evaluate the effectiveness of a variety of behaviorally-informed outreach text messages. The investigators intend to launch the study as a part of UCLA Health's My Action Plan initiative, a UCLA Health primary care outreach quality improvement initiative aimed at encouraging patients to complete their overdue health maintenance measures.

Specifically, the My Action Plan initiative is an outreach effort targeting primary care patients at UCLA who have an outstanding, clinically indicated primary care preventative care gap (e.g., overdue colorectal cancer screening, outstanding diabetes tests). At the beginning of each month, identified UCLA Health primary care patients will be randomized in a 1:1:1:1 ratio to receive one of four text messages informing them that they have an overdue health maintenance measures and urging them to taking action to complete these measures. These text messages will contain a link to their MyChart patient portal account, specifically linking them to a My Action Plan electronic letter that will contain a personalized list of outstanding preventive care items and actionable steps to complete the items.

Within each text-message arm, patients will also be randomized to one of three time slots for getting the message.

The My Action Plan quality improvement initiative is expected to start at the beginning of the 2023 calendar year and continue for a span of at least 12 months. Each month, the initiative targets patients whose birthday falls into that month. The investigators plan to run this randomized clinical trial during four months of the larger QI initiative.

By studying how patients interact with these outreach messages and whether it then translates to them completing their indicated health maintenance measures, the proposed study would provide insightful information on how health systems could optimize electronic patient outreach, narrow the gap in health maintenance measures in primary care, and ultimately improve health on a population level.

Analysis Plan:

* The investigators will utilize patient-level ordinary least squares (OLS) estimation, with statistical inferences based on model-robust standard errors. The primary model term will be indicator variables for arm assignment.
* The analysis will adjust for sex, age, race/ethnicity, indicators for screenings/tests that patients are due for, and whether patients have upcoming primary care appointments. Missing covariate values will be handled by including 'unknown' indicators, along with mean imputation for quantitative covariates.
* The investigators will use this dataset to address two separate research questions.
* Research question 1: The investigators will compare Arm 1 with Arm 2 to test whether more specific or general text message is more likely to improve the outcome measures
* Research question 2: The investigators will compare Arm 3, Arm 4, with Arm 2 to test whether the general intention-oriented message and general action-oriented message can outperform the general text message as well as which of these two messages is better.
* For research question 2, exploratory analyses will investigate heterogeneous treatment effects by patients' baseline motivation (i.e., the extent to which patients seem to have some intentions to get the screenings/tests) in two ways. First, the investigators will use each patient's history of screenings/tests to construct a proxy for their baseline motivation to obtain the due screenings/tests. Specifically, the investigator will calculate, among all the screenings/tests that are included in the My Action Plan Initiative and that a patient was due for in the past few years (exact time window TBD based on data availability), what percentage was completed by the patient (as far as UCLA Health could tell). A higher percentage indicates a higher baseline motivation to get the screenings/tests patients are due for during the study period. Second, the investigators will obtain demographics and medical information that UCLA Health is willing to provide (e.g., gender, age, race/ethnicity, history of cancer and other pre-existing conditions, family cancer history, past adherence to screenings/tests that are included in the My Action Plan Initiative, past receipt of influenza vaccination, frequency of doctor visits; time window of these variables is TBD depending on data availability). With such information, the investigators will train an algorithm to predict patients' baseline motivation level using patients in Arm 2 as the ground truth. Specifically, the investigators will take the aforementioned information about patients in Arm 2 as input, and use whether they complete any of the screenings/visits recommended in the My Action Plan letter within 6 months as the outcome measure. Then the investigators will apply the algorithm to all patients to predict their baseline motivation level. For both approaches, the proxy for baseline motivation (Approach 1) and the predicted baseline motivation level (Approach 2) will be used to analyze the heterogeneous treatment effects of Arms 3 and 4 (vs. Arm 2).
* Additionally the investigators will investigate proxies for whether patients face structural barriers to get screenings/tests as moderators, including socioeconomic factors at the zipcode level, insurance type, proxies for accessibility to healthcare resources such as distance from UCLA Health clinics.
* The investigators will also explore how the effect of text messages varies across the three times of the day when the reminders will be sent.

ELIGIBILITY:
Inclusion Criteria:

1. Empaneled to UCLA Health DOM Primary Care
2. Has at least one overdue health maintenance measure that the My Action Plan initiative focuses on
3. Has an active MyChart status
4. Can accept SMS messages from UCLA Health
5. Has a March, April, May or June Birthday

Exclusion Criteria:

1. Under the age of 18
2. Deceased patients
3. Hospice patients
4. Has opted out electronic communication (bulk messages, email, and/or text)
5. For the final analysis, we will further exclude patients who have scheduled appointments for all screening/tests or completed all screenings/tests prior to the date when they are supposed to receive the text message

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40912 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Opening link within SMS Text message | 1 week after getting the outreach text message
  Percentage of participants across the different arms who click on the link from the outreach message

SECONDARY OUTCOMES:
Opening My Action Plan Letter | 1 week after getting the outreach text message
  Percentage of participants across the different arms who open their personalized My Action Plan letter
Direct scheduling appointment rate | 2 weeks after getting the outreach text message
  Rate of which eligible participants directly schedule an appointment for diabetic retinal exams, diabetes education, or breast cancer screening in order to complete these overdue screening/test(s). These screenings/tests have dedicated appointment resources that people can directly schedule for.
Rate of taking action for one overdue screening/test | 2 weeks after getting the outreach text message
  Rate of which participants schedule an appointment to complete their overdue screening/test or start the online tool for colorectal screening
Completion rate of one screening/test | 6 months after getting the outreach text message
  Rate of completion of at least one screening/test within the observation window

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health Department of Medicine, Quality Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make any individual participant data available.